CLINICAL TRIAL: NCT02119195
Title: Increasing Longevity of Composite Restorations With Defective Margins With Sealants. Controlled Clinical Trial 10 Years Follow-up
Brief Title: Increasing Composite Restorations Sealants
Acronym: SEALCOMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Eduardo Fernandez, Prof., University of Chile
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FOUCH2012/10-3
Record Dates: First submitted 2014-04-09; First posted 2014-04-21 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-04

CONDITIONS: Dental Restoration Failure
Keywords: composite; sealant; longevity
MeSH Terms: interventions — Clinpro Sealant

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- No treatment (No Intervention): The composite resin restorations had marginal defects, but were clinically acceptable, did not receive treatment
- Positive control (No Intervention): Composite resins with alpha value in marginal adaptation criteria
- Intervention (Experimental): For this group, defective areas were acid etched with 35% phosphoric acid for 15 seconds. A resin-based sealant (Clinpro Sealant, 3M ESPE) was applied over the defective area. The sealant was polymerized with a photocuring unit (Curing Light 2500, 3M ESPE) for 40 seconds. Rubber dam isolation was used for this procedure
  Interventions: Procedure: Sealant

INTERVENTIONS:
Procedure: Sealant — resin-based sealant (Clinpro Sealant, 3M ESPE)
  Other Names: Clinpro Sealant; Alpha seal; Prime Dent
  Arms: Intervention

SUMMARY:
A cohort of 20 patients aged 18 to 80 years (mean 28.35 years) of both genres females (65%) and males (35%) with 80 composite restorations were recruited at the Operative Dentistry Clinic at the Dental School of the University of Chile. All participants presented with marginal adaptation clinical features that deviated from the ideal and were rated Bravo according to the modified United States Public Health Service (USPHS) criteria for the sealing group and no treatment group. As a positive control were considered composites with alpha values in marginal adaptation. The protocol was approved by the Institutional Research Ethics Committee of the Dental School at the University of Chile (Project PRI-ODO-0207). All of the patients signed informed-consent forms and completed registration form. The selection criteria are summarized below.

DETAILED DESCRIPTION:
Inclusion Criteria for Allocated groups :

Patients with localized marginal deficiencies (Bravo Ryge Criterial) of composite restorations that were clinically judged to be suitable for sealing according to USPHS criteria.

Patients with more than 20 teeth. Restorations in functional occlusions with an opposing natural tooth. Asymptomatic restored tooth. At least one proximal contact area with a neighbouring tooth. Patients are older than 18 years. Patients who agreed and signed a consent form for participating in the study. Area out of the restoration´s failure is in good condition.

Inclusion Criteria for Positive Control group :

Composite resins with alpha value in adaptation marginal criterial

Exclusion criteria:

Patients with contra-indications for regular dental treatment based on their medical history.

Patients with xerostomia or taking medication that significantly decreased salivary flow.

Patients with a high risk of caries. Patients with psychiatric or physical diseases, which interfered with oral hygiene.

Patients with localized marginal deficiencies > 1 mm. and/or secondary caries adjacent to composite restorations , or major defects 2.2 Treatment Group Criteria Initially, 356 restorations (28 patients) were evaluated and assigned in accordance with the modified USPHS criteria, from which 80 were selected in accordance with the inclusion criteria. Restorations with marginal defects (>0.5mm and <1mm) and/or marginal staining (Bravo) were randomly assigned to the Sealing (n = 20) or no treatment (n = 20) group. The randomization was performed by the Power Analysis and Sample Size System (Excel 2000,Microsoft,SEA, USA).

2.3 Restoration Assessment The quality of the restorations was scored according to the modified USPHS criteria. Two examiners underwent calibration exercises each year (JM and EF). The Cohen's Kappa inter-examiner coefficient was 0.74 at the baseline and 0.87 at ten years. Immediately after the treatment (baseline) and 10 years later, the examiners assessed the restorations independently by direct visual and tactile examination with mouth mirror number 5 and explorer number 23 (Hu Friedy Mfg. Co. Inc., Chicago, IL, USA) and indirectly by radiographic examination (bite wing). The four parameters examined were anatomic form, secondary caries, marginal staining and marginal adaptation. If the difference was recorded between the two examiners, and if they could not reach an agreement, a third clinician, who also underwent the calibration exercises (GM), made the final decision.

2.4 Treatment Groups 2.4.1 Sealing For this group, defective areas were acid etched with 35% phosphoric acid for 15 seconds. A resin-based sealant (Clinpro Sealant, 3M ESPE) was applied over the defective area. The sealant was polymerized with a photocuring unit (Curing Light 2500, 3M ESPE) for 40 seconds. Rubber dam isolation was used for this procedure.

2.4.2 No treatment The composite resin restorations had marginal defects, but were clinically acceptable, did not receive treatment.

2.4.3 Positive control Composite resins with alpha value in marginal adaptation criteria

ELIGIBILITY:
Inclusion Criteria:

* Patients with localized marginal deficiencies (Bravo Ryge Criterial) of composite restorations that were clinically judged to be suitable for sealing according to USPHS criteria.
* Patients with more than 20 teeth.
* Restorations in functional occlusions with an opposing natural tooth.
* Asymptomatic restored tooth.
* At least one proximal contact area with a neighbouring tooth.
* Patients are older than 18 years.
* Patients who agreed and signed a consent form for participating in the study.
* Area out of the restoration´s failure is in good condition.

Inclusion Criteria for Positive Control group :

* Composite resins with alpha value in adaptation marginal criterial

Exclusion Criteria:

* Patients with contra-indications for regular dental treatment based on their medical history.
* Patients with xerostomia or taking medication that significantly decreased salivary flow.
* Patients with a high risk of caries.
* Patients with psychiatric or physical diseases, which interfered with oral hygiene.
* Patients with localized marginal deficiencies > 1 mm. and/or secondary caries adjacent to composite restorations , or major defects

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2003-05; Primary Completion 2003-05 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Changes in quality of restorations | 1 year
  The quality of the restorations was scored according to the modified USPHS criteria. Two examiners underwent calibration exercises each year (JM and EF). Immediately after the treatment (baseline) and 10 years later, the examiners assessed the restorations independently by direct visual and tactile examination with mouth mirror number 5 and explorer number 23 (Hu Friedy Mfg. Co. Inc., Chicago, IL, USA) and indirectly by radiographic examination (bite wing). The four parameters examined were anatomic form, secondary caries, marginal staining and marginal adaptation. If the difference was recorded between the two examiners, and if they could not reach an agreement, a third clinician, who also underwent the calibration exercises (GM), made the final decision.

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Fernández, Prof., Principal Investigator — University of Chile
Locations (1):
- Facultad de Odontología Universidad de Chile, Santiago, Chile

REFERENCES:
- [Result] Moncada GC, Martin J, Fernandez E, Vildosola PG, Caamano C, Caro MJ, Mjor IA, Gordan VV. Alternative treatments for resin-based composite and amalgam restorations with marginal defects: a 12-month clinical trial. Gen Dent. 2006 Sep-Oct;54(5):314-8. PMID 17004564
- [Result] Moncada G, Fernandez E, Martin J, Arancibia C, Mjor IA, Gordan VV. Increasing the longevity of restorations by minimal intervention: a two-year clinical trial. Oper Dent. 2008 May-Jun;33(3):258-64. doi: 10.2341/07-113. PMID 18505215
- [Result] Moncada G, Martin J, Fernandez E, Hempel MC, Mjor IA, Gordan VV. Sealing, refurbishment and repair of Class I and Class II defective restorations: a three-year clinical trial. J Am Dent Assoc. 2009 Apr;140(4):425-32. doi: 10.14219/jada.archive.2009.0191. PMID 19339531
- [Result] Fernandez EM, Martin JA, Angel PA, Mjor IA, Gordan VV, Moncada GA. Survival rate of sealed, refurbished and repaired defective restorations: 4-year follow-up. Braz Dent J. 2011;22(2):134-9. doi: 10.1590/s0103-64402011000200008. PMID 21537587
- [Result] Martin J, Fernandez E, Estay J, Gordan VV, Mjor IA, Moncada G. Minimal invasive treatment for defective restorations: five-year results using sealants. Oper Dent. 2013 Mar-Apr;38(2):125-33. doi: 10.2341/12-062C. Epub 2012 Jul 11. PMID 22788726